CLINICAL TRIAL: NCT03815877
Title: The Effect of Caffeine Ingestion in Prevention of Postoperative Ileus After Caesarean Section: A Randomized Controlled Trial
Brief Title: The Effect of Caffeine Ingestion in Prevention of Postoperative Ileus After Caesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Madonna Gamal Garas Benyamine, DR. MADONNA GAMAL GARAS BENYAMINE, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AinShamsU2018455
Record Dates: First submitted 2018-01-17; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Ileus; Cesarean Section Complications; Caffeine
Keywords: Caffeine; Postoperative Ileus; Caesarean Section

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant
Masking Description: All recruited women will be distributed into two groups according to a computer- generated randomization table. The researcher consecutively will open sequentially numbered, opaque, sealed envelopes containing cards with letters either letter (C) or letter (N), Cards with letter (C) will represent the group who will receive the caffeinated coffee and cards with letter (N) will represent the group who will receive the decaffeinated coffee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (C group receiving caffeinated coffee) (Active Comparator): 100cc coffee at 3, 6 and 9 hours after the Cesarean section
  Interventions: Dietary Supplement: Nescafe Gold ® coffee
- The control group (N group receiving decaffeinated coffee) (Placebo Comparator): 100cc decaf coffee at 3, 6, 9 hours after the Cesarean section
  Interventions: Dietary Supplement: Nescafe Gold DECAF® coffee

INTERVENTIONS:
Dietary Supplement: Nescafe Gold ® coffee — Nescafe Gold ® coffee (5gm per 100cc water containing 170 mg of caffeine) will be used for all the women in the intervention group.
  - patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery.
  Arms: The intervention group (C group receiving caffeinated coffee)
Dietary Supplement: Nescafe Gold DECAF® coffee — Nescafe Gold DECAF coffee (5 gm per 100cc water containing 5-10 mg of caffeine) will be used for all the women in the control group.
  the control group will drink 100cc decaffeinated coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery.
  Arms: The control group (N group receiving decaffeinated coffee)

SUMMARY:
Many trials have been made to prevent paralytic ileus , including administration of prokinetic drugs , early resumption of feeding, gum chewing and adequate pain control. Unfortunately, none of these strategies has been completely successful. Recently the effect of caffeine on prevention of postoperative ileus after caesarian section was researched. That's why this study is designed to determine the efficacy of caffeine in prevention of postoperative ileus after caesarean section.

DETAILED DESCRIPTION:
-Study design: This study will include 600 women undergoing their caesarean section. The study aims will be explained to all women and an informed written consent will be taken. All recruited women will be distributed into two groups according to a computerized randomization table. The researcher consecutively will open sequentially numbered, opaque, sealed envelopes containing cards with letters either letter (C) or letter (N), Cards with letter (C) will represent the group who will receive the caffeinated coffee and cards with letter (N) will represent the group who will receive the decaffeinated coffee

Procedure:

* For all women, the anesthetic used will be Marcaine® Spinal heavy 0.5% and fentanyl and for post-operative pain, ketorolac will be used.
* Through Pfannenstiel incision, transverse lower segment uterine incision is done, with the duration of the surgery not exceeding 90 minutes
* women will not be permitted to drink or eat, except for the drink offered by the researcher, till passing flatus. Early ambulation will be encouraged.
* A stethoscope will be used to detect the first intestinal movement each hour after the surgery. The women will be advised to notify the researcher when they pass both flatus and feces.

Intervention:

* The intervention plan will be performed within the first 24 hours after the surgery.
* Provided by the researcher within 10 minutes, patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery, and the control group will drink 100cc decaffeinated coffee with 1 tea spoon added sugar at the same intervals.
* No other liquid will be allowed till passage of flatus and feces in the first day of surgery.
* Nescafe Gold ® coffee (5gm per 100cc water containing 170 mg of caffeine) will be used for all the women in the intervention group. Nescafe Gold DECAF coffee (5 gm per 100cc water containing 5-10 mg of caffeine) will be used for all the women in the control group.
* Statistical Package:
* Data analysis will be performed by Statistical Package for the Social Science (SPSS) 16.0 using descriptive statistics tools, including mean, standard deviation and figures. A t-test will be used to compare mean values of the two groups. P-values, smaller than 0.05, were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing caesarean section
* Spinal anaesthesia
* Total surgery time less than 90 minutes

Exclusion Criteria:

* Previous complicated abdominal surgery or caesarean section with extensive adhesions requiring extensive dissection or intestinal manipulation.
* Caesarean section complicated by postpartum hemorrhage or in the women who received misoprostol.
* Intraoperative intestinal complications.
* Intraoperative respiratory complication.
* Chronic intestinal diseases: irritable or inflammatory bowel diseases.
* Chronic diarrhea or constipation.
* Using laxatives pre-operatively.
* Known hypersensitivity to caffeine
* Thyroid or hepatic disease.
* Cardiac arrhythmias

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
A change in the number of hours for women to pass flatus for the first time after an elective caesarean section | patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery. The women will be advised to notify the researcher when they pass flatus.
  A change the number of hours for women to pass flatus for the first time after an elective caesarean section

SECONDARY OUTCOMES:
A change in the number of hours for the women to have their first intestinal sound to be heard by a stethoscope after caesarean section | patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery. A stethoscope will be used to detect the first intestinal movement every hour after the surgery
  A change in the number of hours for the women to have their first intestinal sound to be heard by a stethoscope after caesarean section.
A difference in the number of hours for the women to pass stool after caesarean section. | patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery. The women will be advised to notify the researcher when they pass feces.
  A difference in the number of hours for the women to pass stool after caesarean section.
A difference in the number of the women's hospital stay hours after caesarean section | calculating the number of the women's hospital stay hours after caesarean section up to 12 weeks
  A difference in the number of the women's hospital stay hours after caesarean section
Occurrence of postoperative spinal headache | patients will drink 100cc coffee with 1 tea spoon added sugar at 3, 6 and 9 hours after the surgery. The women will be advised to notify the researcher with the occurrence, severity and relief of spinal headache during the hospital stay.
  Occurrence of postoperative spinal headache

CONTACTS AND LOCATIONS:
Overall Officials: AMR NADIM, Study Director — Ain Shams University; REDA GHANEM, Study Director — Ain Shams University; MADONNA BENYAMINE, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Artinyan A, Nunoo-Mensah JW, Balasubramaniam S, Gauderman J, Essani R, Gonzalez-Ruiz C, Kaiser AM, Beart RW Jr. Prolonged postoperative ileus-definition, risk factors, and predictors after surgery. World J Surg. 2008 Jul;32(7):1495-500. doi: 10.1007/s00268-008-9491-2. PMID 18305994
- [Background] Beck DE, Sweeney WB, McCarter MD; Ipamorelin 201 Study Group. Prospective, randomized, controlled, proof-of-concept study of the Ghrelin mimetic ipamorelin for the management of postoperative ileus in bowel resection patients. Int J Colorectal Dis. 2014 Dec;29(12):1527-34. doi: 10.1007/s00384-014-2030-8. Epub 2014 Oct 21. PMID 25331030
- [Background] Bragg D, El-Sharkawy AM, Psaltis E, Maxwell-Armstrong CA, Lobo DN. Postoperative ileus: Recent developments in pathophysiology and management. Clin Nutr. 2015 Jun;34(3):367-76. doi: 10.1016/j.clnu.2015.01.016. Epub 2015 Jan 31. PMID 25819420
- [Background] Brown SR, Cann PA, Read NW. Effect of coffee on distal colon function. Gut. 1990 Apr;31(4):450-3. doi: 10.1136/gut.31.4.450. PMID 2338272
- [Background] Drake TM, Ward AE. Pharmacological management to prevent ileus in major abdominal surgery: a systematic review and meta-analysis. J Gastrointest Surg. 2016 Jun;20(6):1253-64. doi: 10.1007/s11605-016-3140-0. Epub 2016 Apr 12. PMID 27073081
- [Background] Ertas IE, Gungorduk K, Ozdemir A, Solmaz U, Dogan A, Yildirim Y. Influence of gum chewing on postoperative bowel activity after complete staging surgery for gynecological malignancies: a randomized controlled trial. Gynecol Oncol. 2013 Oct;131(1):118-22. doi: 10.1016/j.ygyno.2013.07.098. Epub 2013 Jul 29. PMID 23906657
- [Background] Gungorduk K, Ozdemir IA, Gungorduk O, Gulseren V, Gokcu M, Sanci M. Effects of coffee consumption on gut recovery after surgery of gynecological cancer patients: a randomized controlled trial. Am J Obstet Gynecol. 2017 Feb;216(2):145.e1-145.e7. doi: 10.1016/j.ajog.2016.10.019. Epub 2016 Oct 22. PMID 27780709
- [Background] Holte K, Kehlet H. Postoperative ileus: progress towards effective management. Drugs. 2002;62(18):2603-15. doi: 10.2165/00003495-200262180-00004. PMID 12466000
- [Background] Muller SA, Rahbari NN, Schneider F, Warschkow R, Simon T, von Frankenberg M, Bork U, Weitz J, Schmied BM, Buchler MW. Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy. Br J Surg. 2012 Nov;99(11):1530-8. doi: 10.1002/bjs.8885. Epub 2012 Sep 14. PMID 22987303
- [Background] Rabiepoor S, Yas A, Navaei J, Khalkhali HR. Does coffee affect the bowel function after caesarean section? Eur J Obstet Gynecol Reprod Biol. 2018 Jan;220:96-99. doi: 10.1016/j.ejogrb.2017.07.028. Epub 2017 Aug 4. PMID 29202396
- [Background] Sunil S, Sinha S. Postoperative ileus: a preventable event (Br J Surg 2000; 87: 1480-93). Br J Surg. 2001 Apr;88(4):594-5. doi: 10.1046/j.1365-2168.2001.01787-3.x. No abstract available. PMID 11298633
- [Background] Tan EK, Cornish J, Darzi AW, Tekkis PP. Meta-analysis: Alvimopan vs. placebo in the treatment of post-operative ileus. Aliment Pharmacol Ther. 2007 Jan 1;25(1):47-57. doi: 10.1111/j.1365-2036.2006.03150.x. Epub 2006 Oct 17. PMID 17042776
- [Background] Teoh WH, Shah MK, Mah CL. A randomised controlled trial on beneficial effects of early feeding post-Caesarean delivery under regional anaesthesia. Singapore Med J. 2007 Feb;48(2):152-7. PMID 17304396
- [Background] Toyomasu Y, Mochiki E, Morita H, Ogawa A, Yanai M, Ohno T, Fujii T, Tsutsumi S, Asao T, Kuwano H. Mosapride citrate improves postoperative ileus of patients with colectomy. J Gastrointest Surg. 2011 Aug;15(8):1361-7. doi: 10.1007/s11605-011-1567-x. Epub 2011 May 24. PMID 21607794
- [Background] Zhuang CL, Ye XZ, Zhang CJ, Dong QT, Chen BC, Yu Z. Early versus traditional postoperative oral feeding in patients undergoing elective colorectal surgery: a meta-analysis of randomized clinical trials. Dig Surg. 2013;30(3):225-32. doi: 10.1159/000353136. Epub 2013 Jul 6. PMID 23838894

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03815877/Prot_SAP_000.pdf